CLINICAL TRIAL: NCT03957772
Title: The Efficacy of Extra- Versus Intrafascial Injection for Supraclavicular Brachial Plexus Block: a Randomized Controlled, Single-blinded Trial
Brief Title: The Efficacy of Extra- Versus Intrafascial Injection for Supraclavicular Brachial Plexus Block
Acronym: SUPRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hôpital du Valais (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019 SUPRA
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Upper Extremity Problem
Keywords: upper extremity surgery

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider
Masking Description: The participants and all care providers will be blinded to the patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extrafascial injection (Active Comparator): Extrafascial injection of local anesthetic
  Ultrasound guided supraclavicular plexus block with extrafascial injection of local anesthetic
  Interventions: Procedure: Extrafascial injection
- Intrafascial injection (Experimental): Intrafascial injection of local anesthetic
  Ultrasound guided supraclavicular plexus block with intrafascial injection of local anesthetic
  Interventions: Procedure: Intrafascial injection

INTERVENTIONS:
Procedure: Extrafascial injection — Extrafascial injection of local anaesthetic under ultrasound guidance
  Arms: Extrafascial injection
Procedure: Intrafascial injection — Intrafascial injection of local anaesthetic under ultrasound guidance
  Arms: Intrafascial injection

SUMMARY:
Patients will be randomized to one of two groups:

1. Extrafascial injection group: Ultrasound-guided supraclavicular brachial plexus block with 2 injections of local anaesthetic, deposited at the exterior of the fascial sheath that surrounds the nerves
2. Intrafascial injection group: Ultrasound-guided supraclavicular brachial plexus block with 2 injections of local anaesthetic, deposited at the interior of the fascial sheath that surrounds the nerves

DETAILED DESCRIPTION:
The study will be proposed to all patients undergoing formarm or hand surgery under axillary brachial plexus block. Patients will be randomized to one of two groups.

The first group - extrafascial injection group - will receive an ultrasound-guided supraclavicular brachial plexus block whereby the local anesthetic will be deposited at the exterior of the fascial sheath that surrounds the nerves.

The second group - intrafascial injection group - will receive an ultrasound-guided supraclavicular brachial plexus block whereby the local anesthetic will be deposited at the interior of the fascial sheath that surrounds the nerves.

All patients will receive the same type and amount of local anesthetic: 30 ml of a mixture of ropivacaine 0.5 % + mepivacaine 1 %.

The primary outcome is the rate of hemidiaphragmatic paresis 30 minutes after the block procedure, assessed with ultrasound. Secondary outcomes are: rate of hemidiaphragmatic paresis 2 hours after surgery, assessed with ultrasound, bedside spirometry before the supraclavicular block, 30 minutes after the block and 2 hours after surgery, rate of successful block 30 minutes after the block , duration of sensory and motor block, pain scores at rest and on movement at 24 h postoperatively, cumulative postoperative opioid consumption at 24 hours postoperatively and patient satisfaction with overall anesthetic management.

These outcomes are further defined in the section below.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing forearm or hand surgery under locoregional anesthesia
* ASA physical status I-III

Exclusion Criteria:

* Patient refusal
* ASA physical status IV
* Severe pre-existing lung disease
* Patient unwilling or unable to perform incentive spirometry
* Local anesthetic intolerance or allergy
* Neurological deficit or neuropathy of the arm
* Coagulopathy contraindicating locoregional anesthesia
* Malignancy or infection in the area above the clavicle
* Pregnancy
* Inability to understand the informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Hemidiaphragmatic paresis 30 minutes after the block | 30 minutes after the block
  Rate of hemidiaphragmatic paresis 30 minutes after the block procedure, assessed with ultrasound

SECONDARY OUTCOMES:
Hemidiaphragmatic paresis 2 hours after surgery | 2 hours after surgery
  Rate of hemidiaphragmatic paresis 2 hours after surgery, assessed with ultrasound
Bedside spirometry before the block (baseline) | 30 minutes before the block
  Bedside spirometry before the supraclavicular block
Bedside spirometry after 30 minutes after the block | 30 minutes after the supraclavicular block
  Bedside spirometry after the supraclavicular block
Bedside spirometry 2 hours after surgery | 2 hours after surgery
  Bedside spirometry 2 hours after surgery
Rate of successful block 30 minutes after the block | 30 minutes after the block
  Presence of a surgical block according to a validated composite scale
Block-related side effects | 24 h postoperatively
  paresthesia, dyspnea, Horner's syndrome, hoarseness, hematoma, infection
Pain during block procedure | During block procedure
  Pain score (numeric rating scale, 0-10, with 0=no pain, 10=worst imaginable pain)
Pain at rest and on movement | 24 h postoperatively
  Pain score (numeric rating scale, 0-10, with 0=no pain, 10=worst imaginable pain)
Postoperative opioid consumption | 24 hours postoperatively
  Cumulative postoperative opioid consumption
Patient satisfaction with overall anesthetic management | 24 hours postoperatively
  numeric rating scale, 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Sina Grape, MD, Principal Investigator — Hôpital du Valais
Locations (1):
- Hopital du Valais, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: No
no sharing of any IPD

REFERENCES:
- [Derived] Grape S, Kirkham K, Zemirline N, Bikfalvi A, Albrecht E. Impact of an extrafascial versus intrafascial injection for supraclavicular brachial plexus block on respiratory function: a randomized, controlled, double-blind trial. Reg Anesth Pain Med. 2022 Oct;47(10):604-609. doi: 10.1136/rapm-2022-103634. Epub 2022 Jul 1. PMID 35777931